CLINICAL TRIAL: NCT06896981
Title: Comparison Between the Effects of Low-Dose Semaglutide With Metformin vs. Metformin Alone Over Metabolic Profile in Obese Polycystic Ovary Syndrome: A Phase II Randomized Controlled Trial
Brief Title: Semaglutide in Women With Polycystic Ovary Syndrome and Obesity
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, MA Hasanat, Professor of Endocrinology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.BSMMU/2024/12253-5292
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Polycystic Ovary Syndrome (PCOS) Women; Obesity
Keywords: Polycystic ovary syndrome; Obesity; Semaglutide; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Metformin; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Immediately release metformin 500 mg bd for 12 weeks
  Interventions: Drug: Metformin with Semaglutide
- Metformin and semaglutide (Experimental): Immediately release metformin 500 mg bd for 12 weeks and Inj Semaglutide 0.5 mg once weekly for 12 weeks
  Interventions: Drug: Metformin with Semaglutide

INTERVENTIONS:
Drug: Metformin with Semaglutide — One arm: Metformin 500 mg bd, Other arm: Metformin 500 mg bd + Semaglutide 0.5 mg once weekly

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a common endocrine disorder that is frequently associated with metabolic features, including obesity. Improvement of metabolic manifestations helps in the control of symptoms, including subfertility. Metformin has been commonly used to decrease insulin resistance and weight in PCOS patients suffering from obesity. Glucagon-like peptide (GLP-1) agonist semaglutide is also effective in managing different metabolic features, including obesity and insulin resistance. There is limited data about using a combination of semaglutide and metformin in women with PCOS suffering from obesity. This study aims to compare the metabolic changes after giving a combination of low-dose semaglutide and metformin vs. metformin alone over 12 weeks among women with PCOS and obesity. This open label randomized trial will be conducted in the Department of Endocrinology, Bangabandhu Sheikh Mujib Medical University (BSMMU). After obtaining informed written consent, a total of 30 patients with PCOS and obesity will be enrolled conveniently (sampling) in the study as per inclusion and exclusion criteria from the outdoor, indoor, and PCOS clinic, Endocrinology, BSMMU. Study participants will be divided into two groups randomly by a computerized random number generator (allocation). One study arm will be treated with low-dose subcutaneous semaglutide (0.25 mg/week for 4 weeks followed by 0.5mg per week for 12 weeks) in combination with metformin (500 mg bid). Another study arm will receive monotherapy with metformin (500 mg bid) for treatment. Both arms will receive standard unified lifestyle advices. Patients will be followed every four weeks for clinical data for up to twelve weeks. Laboratory tests will be done at baseline and the final follow-up in an 8 - 12 hours of fasting state. Two mL of blood will be used to measure glucose using the glucose oxidase method on the same day of sample collection. The remaining three mL of blood will be centrifuged, the serum will be separated and analyzed for insulin, TT, SHBG, ALT and lipid profiles on the same day. All the clinical and biochemical information will be documented in a pretested, semi-structured case record form. Recorded data will be entered, edited, and analyzed by SPSS software version 25.0. Data will be expressed as frequencies & percentages (%) for qualitative values and mean & standard deviation (±SD) or median & inter-quartile range (IQR) for quantitative values depending on their distribution. Kaplan Meier Curve will be used to show the comparison between primary outcomes. For quantitative variables, a comparison between two groups will be done using Mann-Whitney U test, and within a group, a paired t-test or Wilcoxon test will be used. For qualitative variables, a comparison between two groups will be tested using Pearson's chi-square test and within the group by the McNemar test. Regression Analysis will be done to correlate between treatment and outcome. Any p-value below 0.05 will be considered statistically significant. Confidentiality will be strictly maintained. Informed written consent will be taken from patients.

DETAILED DESCRIPTION:
Introduction Polycystic ovary syndrome (PCOS) is a prevalent endocrine disorder, impacting approximately 10-20% of women in their reproductive years. The syndrome is typically characterized by reproductive and dermatological manifestations such as irregular menstrual cycles, subfertility, hirsutism, and acne. However, the metabolic components of PCOS, including obesity, hypertension, glucose intolerance, dyslipidemia, and metabolic syndrome, significantly influence the clinical presentation and treatment outcomes of the disease. These metabolic features are primarily associated with insulin resistance and hyperandrogenemia, the key pathological mechanisms of PCOS. Obesity affects about two-thirds of individuals with PCOS and it exacerbates PCOS manifestations, including hyperandrogenism, and decreases fertility rates. It has been demonstrated that the prevalence of PCOS differs across ethnic groups, with higher prevalence reported in South Asian, and lower prevalence in East Asian patients, in comparison to Caucasian women. South Asian is a collective word used to refer to people who originate from the Indian subcontinent (India, Pakistan, Sri Lanka, Bangladesh, and Nepal). These countries are densely populated and, like many regions of the world, also have people who suffer from PCOS. The South Asian population, in general, also exhibits a higher prevalence of insulin resistance and type 2 diabetes, which may increase long-term morbidity among those with PCOS. Weight loss through lifestyle modifications and bariatric surgery has been shown to alleviate all PCOS symptoms, including ovulation improvement, decreased artificial reproductive techniques requirement, and increased pregnancy rate. Resolution of all three diagnostic features of PCOS after lifestyle therapy and bariatric surgery has been demonstrated. Hence, obesity is now considered a secondary cause of PCOS (pseudo-PCOS).

Lifestyle is the cornerstone in the management of PCOS and obesity. According to the American Diabetes Association (ADA), a 5% or greater weight loss can improve metabolic outcomes in obese patients. Metformin, an insulin sensitizer is now an evidence-based treatment option especially those with a body mass index (BMI) at or above 25 kg/m2. Metformin is essentially weight neutral. However, a placebo-controlled double blind randomized controlled trial conducted in our Department showed significant reduction of BMI and waist circumference (WC) over a period of nine months among women with PCOS. Recent studies have demonstrated significant weight reductions in various conditions related to PCOS, including diabetes mellitus (DM), metabolic dysfunction-associated steatotic liver disease, and obstructive sleep apnea, using different types of glucagon-like peptide 1 receptor agonists 1 (GLP1RAs). Another open-label randomized controlled trial from our Department showed more improvement in BMI and insulin resistance (IR) among women with PCOS who were treated with both metformin and liraglutide over twelve weeks than metformin alone. Systematic reviews and meta-analyses have shown significant improvements in weight, waist circumference, and insulin resistance with different GLP1RAs compared to placebo and metformin among women with PCOS. However, these studies primarily included liraglutide and exenatide. There are few studies done on the use of semaglutide in the management of PCOS with obesity.

This study aims to compare the effects of metformin vs. a combination of low-dose semaglutide and metformin on the clinical profile of women with PCOS, providing valuable insights into a potential therapeutic approach for this common endocrine disorder.

Rationale A minimum of 5% weight reduction can ameliorate various symptoms of PCOS, and these improvements continue with further weight loss. However, in most instances, lifestyle modifications alone are insufficient to achieve this. Some patients are intolerant to higher doses of metformin. Low-dose semaglutide combined with a reduced dose of metformin can be an effective synergistic combination of choice for weight loss along with avoidance of side effects. Local semaglutide (non-comparable biologics) is now available in Bangladesh with reduced cost and is frequently practiced in the management of DM and obesity with promising efficacy and tolerability at lower doses. Given that, it can reduce a significant amount of weight in patients with PCOS who are intolerant to high doses of metformin. South Asian patients, who present with more metabolic features, may benefit more from a lower dose of semaglutide, which also has the advantages of lower cost and fewer side effects. Quasi experimental studies already showed some promise. A well designed phase 2 randomized controlled trial in needed for further proof of efficacy, safety and dose response. Therefore, this study aims to compare the effects of a combination of low doses of semaglutide and metformin vs. metformin alone in patients suffering from PCOS and obesity in Bangladeshi women.

Research hypothesis A combination of metformin and subcutaneous low-dose semaglutide improves the metabolic profile better than metformin alone among women with PCOS and obesity.

Research question Does the combination of metformin and subcutaneous low-dose semaglutide improve metabolic outcomes in women with PCOS and obesity better than metformin alone?

Objectives

1. General- To compare the effects in anthropometric and metabolic status (obesity indices, BP, acanthosis nigricans, fasting glucose, fasting insulin, HOMA-IR, lipid profile, and ALT) after treatment by a combination of metformin with semaglutide and metformin alone over 12 weeks among women with PCOS and obesity.
2. Specific-

   1. To compare the clinical and metabolic status at baseline between the groups treated with or without semaglutide
   2. To assess the changes in the clinical and metabolic status from baseline to 12 weeks after treatment within the groups treated with or without semaglutide
   3. To compare the metabolic changes over 12 weeks of treatment between the study groups treated with or without semaglutide
   4. To compare the frequency of participants achieving at least 5% weight loss between the treatment groups with or without semaglutide
3. Others

   1. To compare the side effects between the two treatment groups with or without semaglutide
   2. To compare the changes in FAI between the two treatment groups with or without semaglutide

   Materials and Methods Type of the study Phase II randomized controlled trial Place of study Department of Endocrinology, BSMMU Study period 12 months after approval from IRB Study population Reproductive-aged Bangladeshi women with PCOS and obesity Sample size

   To calculate the sample size for a randomized control trial, the sample size formula for each group in a two-group comparison is as follows:

   n = [(zα/2 + zβ)2 × {p1(1-p1) + p2(1-p2)}] ÷ (p1-p2)2

   Taking the values from a previous similar study,
   * p1 = proportion of incidence in group 1 (5% weight loss in metformin alone group) = 0.25
   * p2 = proportion of incidence in group 2 (5% weight loss in metformin + semaglutide group) = 0.842
   * α = 0.05 (Type I error)
   * β = 0.2 (Type II error, at 90% power)
   * Zα/2 = critical Z value for a 95% confidence level (two-tailed), which is 1.96
   * Zβ = critical Z value for power of 90%, which is 1.28 K = 1 (ratio of sample size between the two groups)

   Calculation of the absolute difference between proportions:

   p1- p2 = 0.25 - 0.842= -0.592

   Calculation of the combined variance:

   p1 × (1 - p1) = 0.25 × (1 - 0.25) = 0.25×0.75 = 0.1875 p2 × (1 - p2) = 0.842 × (1- 0.842) = 0.842×0.158 = 0.133076 p1 × (1 - p1) + p2 × (1 - p2) = 0.1875+0.133076 = 0.320576

   Calculation of the sample size:

   n = {(1.96 + 1.28)2 × 0.320576} ÷ (-0.592)2
   * {(3.24)2 × 0.320576} ÷ 0.350464
   * (10.4976 × 0.320576) ÷ 0.350464 = 3.36527862 ÷ 0.350464 = 9.6023518 ≈ 10 The sample size is 10 for each group. Considering drop-out, at least 15 participants will be included in each group with intention to increase the sample size.

   Sampling method Convenient sampling Data collection technique A semi-structured pretested case record form (CRF) will be used to collect data.

   Inclusion criteria Reproductive-aged women with PCOS diagnosed according to International evidence based guidelines 2023 and obesity

   Exclusion criteria:
   1. Having DM, other significant systemic diseases- chronic kidney disease (eGFR <60mL/minute/ 1.73 m2 BSA), chronic liver disease (ALT >3 × ULN), and heart failure
   2. Patients having PCOS mimicking endocrine disorders (untreated thyroid dysfunctions, hyperprolactinemia, congenital adrenal hyperplasia, Cushing's syndrome, acromegaly, hypothalamic disorder etc.)
   3. Those taking any other weight loss medications (eg., orlistat, liraglutide) within the last 3 months
   4. Those who have undergone bariatric surgery
   5. Any conditions causing weight loss (thyrotoxicosis, Addison's disease, chronic infection, connective tissue disorder, cancer, etc)
   6. Secondary causes of obesity (major mood disorders, steroids, valproate, oral contraceptives, etc)
   7. Contraindications for semaglutide: personal or family history of medullary carcinoma of the thyroid, history of acute pancreatitis, gallbladder disease
   8. Planning for pregnancy or current pregnancy/ lactation

   Study procedure The selection of participants will be based on inclusion and exclusion criteria by convenient sampling.

   1st visit: Informed consent/assent will be taken from patients and will be requested to come fasting on a specific date, time, and place twice a week.

   Related history of the patient will be taken and physical examination will be done. All information will be recorded in a semi-structured case record form.

   A total of 30 PCOS women of reproductive age will be consecutively recruited from the Department of Endocrinology, BSMMU.

   A total of five (05) mL of blood will be collected in the fasting state. Two mL of blood will be used to measure glucose by the glucose oxidase method. The remaining three mL of blood will be centrifuged, the serum will be separated, and insulin, TT, and SHBG will be measured by chemiluminescence immune assay. The lipid profile will be measured by the glycerol phosphate dehydrogenase peroxidase method.

   All the tests will be done on the same day in the Department of Biochemistry & Molecular Biology, BSMMU.

   Allocation of study participants into two intervention groups randomly by a computerized random number generator:

   Group-1: metformin + semaglutide; Group-2: Metformin alone Similar lifestyle advice will be given: 500 Kcal deficient diets + 30 minutes of walking for at least five days a week to all participants.

   Group-1: Immediate-release metformin- 500 mg od in 1st and 2nd week, then 500 mg bd in 3rd and 4th week, then 500 mg bd for further 12 weeks will be given. Semaglutide 0.25 mg sc once weekly for 4 weeks, then if tolerated, will be titrated up to 0.5mg sc and continued for 12 weeks.

   Group-2: Immediate-release metformin- 500 mg od in 1st 2 weeks, then 500 mg bd in 3rd and 4th weeks, then if tolerated, 500 mg bd will be continued for another 12 weeks.
   1. st follow-up after 4 weeks: Assessment of clinical profile, compliance with drug, and side-effects.

      If patients can tolerate:

      Group-1: Continuation of 1000 mg/day of metformin and increase the dose of semaglutide of 0.5 mg sc once weekly for the next 12 weeks Group-2: Continuation of 1000 mg/day of metformin for the next 12 weeks. If patients cannot tolerate it: Reduced doses will be used for the next 12 weeks.
   2. nd follow-up after 8 weeks: Assessment of clinical profile, measurement of Weight, WC, HC, BP, compliance with drug, and side-effects.

      If patients can tolerate:

      Group-1: Continuation of 1000 mg/day of metformin and 0.5 mg of semaglutide sc once weekly for the next 8 weeks Group-2: Continuation of 1000 mg/day of metformin for the next 8 weeks. If patients cannot tolerate: Reduced dose will be used for the next 8 weeks.
   3. rd follow-up after 12 weeks: Assessment of clinical profile, measurement of Weight, WC, HC, BP, compliance with drug, and side-effects.

   If patients can tolerate:

   Group-1: Continuation of 1000 mg/day of metformin and 0.5 mg of semaglutide sc once weekly for the next 4 weeks Group-2: Continuation of 1000 mg/day of metformin for the next 4 weeks. If patients cannot tolerate: Reduced dose will be used for the next 4 weeks.

   Final (4th follow-up visit) after 16 weeks:

   Assessment of clinical profile, measurement of weight, WC, HC, BP compliance with drug and side-effects.

   Again about five (05) mL of blood will be collected in the fasting state. Two mL of blood will be used to measure glucose using the glucose oxidase method on the same day of sample collection. The remaining three mL of blood will be centrifuged, the serum will be separated and analyzed for insulin, TT, SHBG, ALT and lipid profiles on the same day.

   Outcome variables

   Primary endpoints:
   * Weight loss of at least ≥ 5% from baseline after 16 weeks
   * Body mass index
   * Waist circumference
   * Hip circumference
   * Blood pressure
   * Acanthosis nigricans
   * Fasting plasma glucose
   * Fasting insulin
   * Homeostasis model of insulin resistance (HOMA-IR)
   * Lipid Profile

   Secondary endpoints:
   * Total testosterone
   * Sex hormone-binding globulin
   * Free androgen index
   * ALT

   Operational definitions:

   PCOS: PCOS will be diagnosed based on gynecological age Gynecological age ≥8 years: any two of the three following criteria
   * Ovulatory dysfunction is defined by an irregular menstrual cycle
   * Clinical and/or biochemical hyperandrogenism
   * Polycystic ovary morphology by ultrasonography Gynecological age: 1 - 7 years- Both two criteria
   * Ovulatory dysfunction is defined by an irregular menstrual cycle
   * Clinical and/or biochemical hyperandrogenism

   Similar diseases that will be excluded are:
   * Hypothyroidism: clinically and biochemically
   * Hyperprolactinemia: clinically and biochemically
   * Congenital adrenal hyperplasia: Clinically and biochemically
   * Androgen-producing tumor: clinically and biochemically if applicable
   * Acromegaly: Clinically

   Irregular menstrual cycle:

   Irregular menstrual cycles will be defined as:

   • Primary amenorrhoea by age 15 or >3 years post thelarche
   * 1-year post menarche >90 days for any 1-cycle
   * 1 to <3 years post menarche: <21 or >45 days
   * 3 years post menarche to perimenopause: <21 or >35 days or <8 cycles per year When irregular menstrual cycles are present, a diagnosis of PCOS should be considered and assessed according to these PCOS Guidelines Reproductive age: One year after menarche up to perimenopause Obesity: Obesity will be defined by a BMI of ≥27.5 kg/m2 for adults and ≥95th percentile for age and sex for adolescents.

   Polycystic ovarian morphology: Any ovarian volume ≥10 mL or any ovary containing follicle no. (2-9 mm) per section ≥10

   Clinical hyperandrogenism:

   Clinical hyperandrogenism will be defined by the presence of significant hirsutism measured by a modified Ferriman-Gallwey (mFG) score. As there is no population-specific data, the investigators will use the cut-off score of 6 to categorize it as clinical hyperandrogenism.

   Biochemical hyperandrogenism (hyperandrogenemia):

   As there is no population-specific data to define biochemical hyperandrogenism, the investigators will use total testosterone (TT) >46 ng/dL and/or a free androgen index (FAI) ≥5% as a definition of biochemical hyperandrogenism.

   Metformin: Immediate release metformin 500mg from single brand will be used. Low-dose semaglutide: 0.5 mg subcutaneous semaglutide per week

   1 prefilled syringe semaglutide 0.5mg (non-comparable biologics) from single local brand will be used.

   Lifestyle intervention: An energy restricted diet (500 kcal/day reduction) along with at least 30 min of moderate intensity physical activity daily will be recommended to women fulfilling the inclusion criteria.

   Metabolic profile: It includes clinical and biochemical features- Clinical: Weight, BMI, WC, HC, BP, and acanthosis nigricans. Biochemical: FPG, fasting insulin, HOMA-IR, lipid profile, and ALT.

   Others:
   * Central obesity: WC ≥80 cm
   * Glycemic status: According to ADA 2024 guideline
   * Insulin resistance: HOMA-IR ≥2.6, calculated as HOMA-IR = [Fasting insulin (µIU/ml) × Fasting Blood Glucose (mmol/ml)] ÷ 22.5
   * Dyslipidemia: TG ≥150mg/dL and/or HDL Cholesterol <50mg/dL
   * Metabolic dysfunction associated steatohepatitis (MASH): ALT >25 U/L

   Physical measurements:

   Height:

   After removing footwear and headgear, the participants will be asked to stand against a stadiometer with feet together, heels touching the backboard with straight knees, and to look straight ahead maintaining the Frankfurt line. Height will be measured in centimeters (cm) at the exact point to the nearest mm during inspiration with stand tall.

   Weight:

   After placing a digital weighing scale on a flat and firm surface, the participants will be requested to step onto the scale with one foot on each side of the scale after removing footwear, socks, belt, mobile, wallet, etc. Weight will be recorded in kilogram (kg) while the patient remains still with face forward and arms placed on both sides of the trunk.

   BMI (kg/m2):

   BMI of the subjects will be calculated using standard formula, BMI=Weight (kg) / Height (m)2.

   Waist circumference (WC):

   Waist circumference will be measured by a constant tension tape wrapping it around the midpoint between the last palpable rib and the top of the hip bone by keeping it snug while the participant remains standing with weight evenly distributed on both feet, keeping arms relaxed in both sides and during expiration. Reading will be taken to the nearest 0.1 cm.

   Hip circumference (HC):

   Hip circumference will be measured over light clothing in a private area at the maximum circumference over the buttocks with the arms relaxed on both sides and weight evenly distributed on both feet. Measurement will be taken at the level of the tape to the nearest 0.1 cm.

   Blood pressure (BP):

   BP will be measured by sitting quietly in a chair (feet on the floor and back supported, legs uncrossed) for 15 minutes with the arm supported on a table in an empty bladder using a well-calibrated and validated aneroid sphygmomanometer with an appropriate size cuff (bladder encircles 80% of the arm) placed on the patient's upper arm at the level of the right atrium (the midpoint of the sternum) with lower band positioned 2 cm above the elbow. The patient should not have coffee before or during the measurements, and should not talk during the measurements. A stethoscope diaphragm will be used for auscultatory readings. SBP and DBP will be recorded as the onset of the first Korotkoff sound and the disappearance of all Korotkoff sounds, respectively, using the nearest even number. BP will be measured in both arms. Another two measurements will be made at least after three minutes in the arm with the highest measurement. The mean of the last two measurements will be used for systolic and diastolic blood pressure.

   Number of menstruation:

   The total number of spontaneous menstruation within 12 weeks of treatment will be counted.

   Analytic Methods:

   Fasting insulin: It will be measured by chemiluminescence immunoassay (Advia Centaur, Siemens) in the Department of Biochemistry, BSMMU.

   Total testosterone: It will be measured by chemiluminescence immunoassay (ADVIA Centaur CP system) in the Department of Biochemistry, BSMMU.

   Sex hormone binding globulin (SHBG): It will be measured by chemiluminescence immunoassay (ADVIA Centaur CP system).

   Lipid profile: It will be measured by the glycerol phosphate dehydrogenase peroxidase method in the Department of Biochemistry, BSMMU.

   Fasting plasma glucose: Plasma glucose will be analyzed using Dimension EXL 200 Integrated Chemistry System (Siemens, Germany) by glucose-oxidase method in the Department of Biochemistry, BSMMU)

   Data processing and analysis:

   Data from the study will be analyzed using computer-based SPSS Program version 25 (Intel Corporation).

   Statistical methods:

   Data will be expressed as frequencies and percentages (%) for qualitative values and mean and standard deviation (±SD) or median and inter-quartile range (IQR) for quantitative values depending on their distribution. Kaplan Meier Curve will be used to show the comparison between primary outcomes. For quantitative variables, a comparison between two groups will be done using Mann-Whitney U test, and within a group, a paired t-test or Wilcoxon test will be used. For qualitative variables, a comparison between two groups will be tested using Pearson's chi-square test and within the group by the McNemar test. Regression Analysis will be done to correlate between treatment and outcome. Any p-value below 0.05 will be considered statistically significant. Results will be analyzed using intention to treat protocol.

   The study flowchart:

   PCOS patients with obesity in the PCOS clinic, Endocrinology, BSMMU ↓ Inclusion and exclusion criteria + Consent/Assent ↓
   1. st (baseline) visit Weight, height, WC, HC, BP and PCOS-related histories Fasting blood- glucose, insulin, total testosterone, SHBG, ALT and lipid profiles Initiation of drugs + lifestyle management

      ↓
   2. nd visit (after 4 weeks of initial dose) Weight, WC, HC, BP, compliance, side effects, lifestyle Increase the dose of the combination of semaglutide+ metformin or metformin alone to maintenance dose if the initial dose is tolerated

      ↓
   3. rd visit (after 8 weeks of initial dose) Weight, WC, HC, BP, compliance, side effects, lifestyle Continue maintenance dose if the initial dose is tolerated

      ↓
   4. th visit (after 12 weeks of initial dose) Weight, WC, HC, BP, compliance, side effects, lifestyle Continue maintenance dose if the initial dose is tolerated

      ↓
   5. th visit (after 16 weeks of initial dose) Weight, height, WC, HC, BP, compliance, side effects Fasting blood- glucose, insulin, total testosterone, SHBG, ALT and lipid profiles ↓ Data entry, analysis, report writing ↓ Thesis submission

   Quality of assay of laboratory variables The investigators will calibrate the weight machine and sphygmomanometer periodically. The same machines will be used for all the visits. Blood samples will be collected and assayed in a concerned laboratory. Reports will be immediately collected and preserved in the raw data sheet.

   Time table Activity Months

   1 2 - 9 10 11 12 Finalization of protocol Data collection, follow-up, and laboratory analysis Data entry Data editing and analysis Report writing, submission

ELIGIBILITY:
Inclusion Criteria:

Reproductive-aged women with PCOS diagnosed according to International evidence based guidelines 2023 and obesity

Exclusion Criteria:

1. Having DM, other significant systemic diseases- chronic kidney disease (eGFR <60mL/minute/ 1.73 m2 BSA), chronic liver disease (ALT >3 × ULN), and heart failure
2. Patients having PCOS mimicking endocrine disorders (untreated thyroid dysfunctions, hyperprolactinemia, congenital adrenal hyperplasia, Cushing's syndrome, acromegaly, hypothalamic disorder etc.)
3. Those taking any other weight loss medications (eg., orlistat, liraglutide) within the last 3 months
4. Those who have undergone bariatric surgery
5. Any conditions causing weight loss (thyrotoxicosis, Addison's disease, chronic infection, connective tissue disorder, cancer, etc)
6. Secondary causes of obesity (major mood disorders, steroids, valproate, oral contraceptives, etc)
7. Contraindications for semaglutide: personal or family history of medullary carcinoma of the thyroid, history of acute pancreatitis, gallbladder disease
8. Planning for pregnancy or current pregnancy/ lactation

Ages: 10 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 weeks
  in Kg, at least 5% weight loss
Body mass index | 12 weeks
  Kg per meter square
Waist circumference | 12 weeks
  Centimeter
Hip circumference | 12 weeks
  Centimeter
Blood pressure | 12 weeks
  mm of Hg
Acanthosis nigricans | 12 weeks
  Present or absent
Fasting plasma glucose | 12 weeks
  mmol/L
Fasting insulin | 12 weeks
  micro international unit per mL
Homeostasis model assessment of insulin resistance | 12 weeks
  Using formula provided by Mathew's et al. (1985)
Total cholesterol | 12 weeks
  mg/dL
HDL-cholesterol | 12 weeks
  mg/dL
LDL-cholesterol | 12 weeks
  mg/dL
Triglyceride | 12 weeks
  mg/dL

SECONDARY OUTCOMES:
Total testosterone | 12 weeks
  ng/dL
Sex hormone binding globulin | 12 weeks
  nmol/L
Free androgen index | 12 weeks
  in %
Alanine amino transferase | 12 weeks
  U/L

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abul Hasanat, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Department of Endocrinology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication